CLINICAL TRIAL: NCT03365414
Title: A Double Blind Randomized Controlled Crossover Study to Systematically Assess the Efficacy and Safety of Intravenous Albumin Infusions in Severe Postural Orthostatic Tachycardia Syndrome
Brief Title: A Study to Systematically Assess the Efficacy and Safety of Intravenous Albumin Infusions in Severe POTS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawal of support of product for trial
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ZS-POTS-2017
Record Dates: First submitted 2017-08-24; First posted 2017-12-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-07

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: Postural Orthostatic Tachycardia Syndrome; POTS; Syncope; Vasovagal; Hypotension; Tachycardia
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Syncope; Hypotension; Tachycardia | interventions — Albumins; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Phase I (albumin or normal saline): 4 weeks -> washout/crossover: 4 weeks ->Phase II(albumin or normal saline, whichever wasn't administered in phase I): 4 weeks
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase I (Other): Placebo ( Normal Saline 0.9% Infusion Solution Bag) or active comparator (Albumin (Human) 5%, USP)
  Interventions: Biological: Albumin (Human) 5%, USP; Drug: Normal Saline 0.9% Infusion Solution Bag
- Phase II (Other): Placebo ( Normal Saline 0.9% Infusion Solution Bag) or active comparator (Albumin (Human) 5%, USP), whichever was not not administered in Phase I
  Interventions: Biological: Albumin (Human) 5%, USP; Drug: Normal Saline 0.9% Infusion Solution Bag

INTERVENTIONS:
Biological: Albumin (Human) 5%, USP — Albumin (Human) 5%, USP. Intravenous Solution. Plasma Substitute/Blood Derivative
Drug: Normal Saline 0.9% Infusion Solution Bag — Placebo Normal Saline 0.9% Infusion Solution Bag.
  Other Names: sodium chloride 0.9% infusion solution bag

SUMMARY:
POTS is a relatively common condition that affects millions of patients around the globe. It has an estimated prevalence of 170/100,000 with approximately 80% of patients being women of childbearing age. POTS is characterized by an excessive heart rate increase on assuming an upright posture, either standing or even sitting and leading to disabling palpitations, light-headedness, and even in syncope in severe cases. More than 95% patients with POTS have pronounced cardiovascular deconditioning and show marked exercise intolerance. The severity of POTS is variable. In mild cases the affected patient may continue with routine activities with minimal limitations. Severe form of the disease precludes most normal life activities, such as sitting upright, walking or standing to perform even basic house chores. An estimated 40% of patients with POTS have a resistant form of the condition that is nonresponsive or mildly responsive to all treatments resulting in continued functional limitations in the long term.

Many of the currently available treatments in POTS are geared towards increasing blood pressure. These include compression stockings, increased daily fluid intake and increased salt ingestion. Saline infusions may be helpful in certain patients in the short term, though many do not respond. The effectiveness of medications varies greatly, with many patient failing to improve.

A small series of clinical patients suffering from severe POTS have shown robust response to weekly albumin therapy, which supports the hypothesis that periodic albumin infusions will provide significant and sustained symptomatic relief to patients with severe POTS.

This pilot study will explore the effectiveness of albumin infusions as a treatment for POTS. Eligible patients will receive weekly intravenous infusions of 5% Albumin or Saline in a double blinded fashion for 4 weeks and will crossover to the other infusion for 4 weeks after an intervening 4-week washout period. The participants will be required to maintain a daily diary of their symptoms during the screening, the study and washout periods. Any possible adverse effects as the result of infusions will be documented. Outcome measures will be quantified and validated at the end of each study period and the percentage reduction of tachycardia will be determined at the completion of each study arm.

DETAILED DESCRIPTION:
Purpose

To assess the efficacy and safety of intravenous 5% albumin infusions in severe Postural Orthostatic Tachycardia Syndrome (POTS).

Hypothesis

Periodic albumin infusions will be effective in treating patients with severe Postural Orthostatic Tachycardia Syndrome (POTS)

Justification

POTS is characterized by an excessive increase in heart rate and light-headedness on assuming an upright posture, standing or sitting that at times culminates in syncope. Most symptoms of POTS result from marked cardiovascular deconditioning and activation of sympathetic responses due to cerebral hypoperfusion. Plasma volume expanding therapies are one of the mainstays of treatment. Saline infusions in patients with severe orthostatic intolerance lead to rapid but transient symptomatic improvement lasting several hours. Human albumin infusions are used for plasma volume replacement/expansion and have been shown to significantly improve cerebral blood flow. A small subset of patients suffering from severe POTS have shown robust response to weekly albumin therapy, supporting the investigator's hypothesis that periodic albumin infusions will provide significant and sustained symptomatic relief to patients with severe POTS. This would increase their orthostatic tolerance and improve functional capacity without the limitations and side effects associated with other therapies.

Objectives

Primary Objective:

Measured change in the severity of orthostatic intolerance assessed by the Orthostatic Symptom Grading Scale (OSGS) scores at 4 weeks in each arm of the study.

Secondary Objectives:

Measured changes in Patient-Reported Outcomes Measurement Information System, Health Assessment Questionnaire (HAQ -20) from baseline to end of study.

Degree of improvement from baseline in the severity of tachycardia and pulse pressure on a 10-minute HUTT.

Exercise Testing: Change in maximal exercise capacity of the patients from baseline using peak oxygen consumption (VO2).

Research Method/Procedures

Study Duration: 2 years

Subject Duration: 16 weeks; 15 visits (+2 optional)

This is a pilot study with a randomized double blind, controlled, and cross over design.

Fifteen patients with severe neuropathic form of primary POTS will be enrolled from the University of Alberta Hospital (UAH) Autonomic Clinic during the two-year study period.

Eligible patients will receive weekly intravenous infusions of 5% Albumin or Saline in a double blinded fashion for 4 weeks and will crossover to the other infusion for 4 weeks after an intervening 4-week washout period.

The participants will be required to maintain a daily diary of their symptoms during the screening, the study and washout periods. Any possible adverse effects as the result of infusions will be documented.

Outcome measures will be quantified using validated symptom scales at the end of each study period and the percentage reduction of tachycardia from baseline on tilt table test done within three days of completion of each study arm.

Subjects will be randomized to one of two treatment arms: one arm will receive 5% albumin at a dose of 1 gm/kg to be given weekly for 4 weeks and the other arm will receive an equal amount on a volume basis of Saline weekly for 4 weeks. At the end of this treatment period the subjects will undergo a 4-week washout period followed by opposite treatment arm from the first study period. In this protocol each patient will serve as their own control.

Study Procedures

1. Physical/Neurologic Examination

   All patients will undergo detailed a physical/neurological examination and laboratory testing at the time of enrolment and during the study.
2. Cardiac Workup

   All participants will have had an ECG and an echocardiogram. If not one will be done prior to enrolment.
3. Autonomic Testing

Patients will also undergo detailed autonomic testing as per Mayo Clinic Protocols at baseline, which will include the following tests:

i. Quantitative Sudomotor Axon Reflex Test (Sweat testing) will be done to rule out autonomic failure as a cause of orthostatic intolerance. An abnormal sweat test in the foot/leg is seen in neuropathic form of POTS and suggest postganglionic sympathetic Sudomotor involvement. Sweat responses will be recorded from four consistent sites (left forearm, proximal lateral leg, medial distal leg, and proximal foot). Test interpretation will involve comparison of observed sweat volumes (in nl/min) with age- and gender-based norms.

ii. Cardiovagal (Parasympathetic) Testing: Parasympathetic (cardiovagal) function will be assessed by measuring heart rate variability (HRV) during deep breathing (DB), Valsalva Maneuver (VM) and HUTT and the responses compared to age based normal. Briefly, during the DB test the patient will perform deep inspirations and expirations paced to an oscillating light emitting diode (LED). Beat-to-beat R-R intervals will be recorded during each effort and the mean HRV range determined by averaging the largest R-R differences for five consecutive cycles. During the VM, patients will blow into a tube at a constant pressure for 15 seconds while supine. Valsalva ratio (VR) will be calculated by dividing the maximum HR by lowest HR occurring within 40 seconds after VM. Finally, during HUTT the 30:15 ratio will be calculated by dividing R-R interval at 30 secs to the R-R interval at 15 secs while inclined.

iii. HUTT will be done at baseline for confirmation of diagnosis and to assess severity of POTS i.e. orthostatic tachycardia, pulse pressure reduction, neurocardiogenic syncope, and within three days of the end of each arm of the study. Heart rate will be recorded continuously with a 3-lead ECG. After baseline recording for 2-5 minutes, patients will be tilted to an angle of 70 degrees for 10 minutes after which patients will be reclined back to supine position for another 5 minutes. The blood pressures will be manually recorded from the opposite arm at 30 seconds, 1 minute, 2 minute, 5 minute, 7 minute and 10 minutes. Symptoms and signs of presyncope will be monitored and recorded throughout the duration of test. HUTT will also be performed at the end of each phase and at end of study (for a study total of four times) to assess efficacy.

d. Exercise Tolerance:

The physical/exercise endurance of the study subjects will be assessed by an exercise physiologist/rehabilitation specialist at baseline and the end to study to assess the effect of intervention on the participants' physical abilities. VO2max will be calculated using standard protocols - measured VO2max (ml/kg/minute) divided by predicted VO2max multiplied by 100.

e. Laboratory Investigations

Laboratory Investigations will be performed during the study visits as shown:

Serum albumin, electrolytes, complete blood count (CBC), d-dimer levels at baseline and every two weeks (to assess hemolysis, volume overload etc.) Supine and standing plasma catecholamine levels at baseline and end of study (to assess sympathetic tone) 24-hour urinary sodium excretion at baseline, mid-point (2weeks) and end of each arm.

- Baseline serum pregnancy test in women.

f. Patient Diaries

Patients will be asked to maintain a daily diary of their symptoms using the OSGS and PHAQ -20 scales, and sleep diaries during the screening and the study periods. Patients will record a twice-daily dairy of supine and orthostatic blood pressures to assess the incidence of any orthostatic hypertension using provided blood pressure monitors. Any possible adverse effects associated with albumin infusions as reported by the study participants or infusion nurses will be noted.

Plan for Data Analysis

Data analysis will be procured through collaboration with Epidemiology Coordinating and Research Centre (EPICORE) at University of Alberta.

The null hypothesis is that the primary outcome measure i.e. OSGS scores at baseline would not be statistically different at the end of study period in the active arm of the study.

For the primary statistical analysis, we will use a paired t-test to compare the OSGS scores at baseline and at 4 weeks in each arm of the study. Secondary analyses will be performed with paired t-test comparing the scores on HAQ-20 scales and degree of tachycardia at same time points. Repeated measures analysis of variance (ANOVA) will be used to compare functional and sleep scores in patients' diaries over the study period. Probability values <.05 will be considered statistically significant, and all tests will be 2-tailed.

Sample size calculation: Number of subjects needed for this study with a power of 0.8, an effect size of 0.7 (from pilot data) and a significance level of .05 is 15. With an estimated dropout rate of 15% (2 patients) the total number of subjects required is 17.

Study Outcome/Duration Rationale: The duration of each arm of the study and outcome measures were determined based on the following observations:

1. Preliminary results indicate that patients start showing symptomatic improvement within few weeks of albumin infusions. The four-week duration for each study arm should be able to discern the differences in clinical benefit between the two infusions.
2. Considering the albumin half-life, a four-week washout period week should allow complete return to baseline without any residual effects from the preceding infusion.
3. Many studies in POTS have used transient changes in cardiovascular parameters i.e. tachycardia, stroke volume etc. immediately after administration of the study drug as surrogate markers of improvement in POTS. These biological markers alone do not necessarily reflect clinical benefit, are one-dimensional and are confounded by a number of physiologic variables. Nevertheless, the degree of improvement in orthostatic tachycardia on tilt table testing has been included as a secondary outcome measure.
4. The primary and secondary end points are geared towards global assessment that incorporate the patients' symptoms and impact of intervention on overall functional scores and orthostatic intolerance over a sustained period. These are unarguably more robust and reflective of the true clinical status.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ages between 18 to 69 years
2. Disease duration of >12 months
3. Diagnosis of idiopathic POTS confirmed by absolute heart rate increase to >120 beats/minute or increase by >30 beats/minute from baseline within 10 minutes on HUTT without orthostatic hypotension (i.e. drop in systolic BP >30mm of Hg) Plus, • Tachycardia, associated with symptoms of orthostatic intolerance (light-headedness, palpitations, chest pain, nausea, visual blurring, sweating, limb paresthesias)

1. Abnormal sweat testing in the leg/foot (to confirm neuropathic POTS) 2. Severe disease manifestations defined as meeting all three of the following criteria:

1. Severe orthostatic intolerance - Orthostatic Symptoms Grading Scale (OSGS) Score >12
2. Severe symptoms that preclude activities of daily living i.e. Patient-Reported Outcomes Measurement Information System, Health Assessment Questionnaire (PHAQ 20) score >36
3. Lack or limited response to an adequate trial (8 weeks' duration) of at least two of the following standard treatment modalities for POTS including

i. Increased daily intake of salt & water ii. Midodrine iii. Fludrocortisone iv. Beta blockers v. Selective Serotonin Reuptake Inhibitors vi. Desmopressin

Exclusion Criteria:

1. Orthostatic hypotension - a decline of 30mm Hg or more in systolic blood pressure or 20mm Hg or more in mean blood pressure within 3 minutes of standing or head-up tilt.
2. Abnormal ECG or echocardiogram.
3. Recent history (<1 month) of protracted diarrhea or vomiting or hospitalization.
4. History of significant psychiatric or eating disorders.
5. Pregnancy or lactation.
6. History of allergic reactions to human albumin.
7. Patients on diuretic, laxative or antihypertensive medications (except beta blockers)
8. Systemic illness affecting autonomic function (pheochromocytoma, congestive heart failure, hypertension, renal or hepatic disease, severe anemia, alcoholism, malignant neoplasm, diabetes, hypothyroidism, or stroke).
9. Presence of any secondary cause of POTS - amyloidosis, sarcoidosis, alcoholism, lupus, Sjögren's syndrome, chemotherapy, and heavy metal poisoning.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Severity of Orthostatic Intolerance | Change in Orthostatic Symptom Grading Scale (OSGS) scores from baseline to end of first arm (1-4 weeks), from end of washout (5-8 weeks) to end of second arm (9-12 weeks) and at end of study (16 week duration).
  Self-reported severity of orthostatic intolerance assessed by the Orthostatic Symptom Grading Scale (OSGS) scores. Recorded daily. Each item is scored 0-4 (0= lowest severity; 4=greatest severity), yielding a total between 0 and 25.

SECONDARY OUTCOMES:
Disability Assessment | Weekly through study completion, 16 week duration
  The Health Assessment Questionnaire (HAQ) score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. For each of the categories, participants reported the amount of difficulty they had in performing 2 or 3 specific subcategory items. The standard disability score is calculated from the 8 categories by dividing the sum of the individual categories by the number of categories answered, yielding a score from 0 (without any difficulty) to 3 (unable to do).
Degree of cardiovascular improvement - Heart rate | Changes in heart rate (BPM) from baseline to end of first arm (1-4 weeks), from end of washout (5-8 weeks) to end of second arm (9-12 weeks) and at end of study (16 week duration).
  Degree of improvement from baseline in the severity of tachycardia (beats per minute) on a 10-minute head up tilt table test (HUTT). The tilt table test will be performed at baseline and at the end-points of each arm of the study to measure degree of heart rate increment and pulse pressure reduction within 10 minutes of assuming an upright posture.
Degree of cardiovascular improvement - Pulse | Changes in blood pressure (mm Hg) from baseline to end of first arm (1-4 weeks), from end of washout (5-8 weeks) to end of second arm (9-12 weeks) and at end of study (16 week duration).
  Degree of improvement from baseline in the pulse pressure (mm Hg) on a 10-minute head up tilt table test (HUTT). The tilt table test will be performed at baseline and at the end-points of each arm of the study to measure degree of heart rate increment and pulse pressure reduction within 10 minutes of assuming an upright posture.
Change in maximal exercise capacity - Cardiopulmonary exercise testing | Changes in aerobic capacity between baseline and end of first arm (1-4 weeks), and end of washout (5-8 weeks) to end of second arm (9-12 weeks). Follow-up data at end of study (16 week duration).
  Cardiopulmonary exercise testing (CPX) using breath by breath gas-analysis measures variables related to cardiorespiratory function, including expiratory ventilation and pulmonary gas exchange (oxygen uptake (VO2) and carbon dioxide (VCO2).The standard expression of aerobic working capacity is the maximum VO2.
  VO2 max reached during a symptom-limited incremental CPX protocol is commonly expressed as O2 per kg-1 per min -1.
Change in maximal exercise capacity - Electrocardiogram | Changes in aerobic capacity between baseline and end of first arm (1-4 weeks), and end of washout (5-8 weeks) to end of second arm (9-12 weeks). Follow-up data at end of study (16 week duration).
  Electrocardiogram (ECG) measures allows for quantitatively linking metabolic, cardiovascular and pulmonary responses to exercise.
Change in maximal exercise capacity - Heart rate | Changes in aerobic capacity between baseline and end of first arm (1-4 weeks), and end of washout (5-8 weeks) to end of second arm (9-12 weeks). Follow-up data at end of study (16 week duration).
  Pulse measures allows for quantitatively linking metabolic, cardiovascular and pulmonary responses to exercise.
Change in maximal exercise capacity - Blood Pressure | Changes in aerobic capacity between baseline and end of first arm (1-4 weeks), and end of washout (5-8 weeks) to end of second arm (9-12 weeks). Follow-up data at end of study (16 week duration).
  Blood pressure measures allows for quantitatively linking metabolic, cardiovascular and pulmonary responses to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Zaeem Siddiqi, MD PhD, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) available with other researchers.